CLINICAL TRIAL: NCT03499301
Title: Description of Chronic Pain in Emergencies Room and Medical Care Modalities
Acronym: CHRODOLURG
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2017/15
Record Dates: First submitted 2018-03-20; First posted 2018-04-17 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2018-03

CONDITIONS: Chronic Pain; Emergency Department
Keywords: Chronic pain; Emergency; Satisfaction
MeSH Terms: conditions — Chronic Pain; Emergencies; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic pain: Patients with chronic pain when arrived to emergency room.
- No chronic pain: Patients without chronic pain when arrived to emergency room.

SUMMARY:
The rate of patients with chronic pain (CP) is 40% in patients with acute pain in emergency department (ED). Patients with CP come more frequently to ED than patients without CP. Reasons for their visit to ED are often in relation with this CP. Few studies have been interested to management modalities of these patients in ED. The investigators are going to realize a prospective observational study in one center. The hypothesis is that patients with chronic pain are less satisfied of ED management that patients without CP.

DETAILED DESCRIPTION:
Chronic pain is defined by a daily pain since more than 3 months. CP is different of acute pain because of their mechanisms, treatments and therapeutic objectives. CP is associated with an alteration of quality of life with psychological, social and economic consequences. The prevalence of CP in France is 15%. In ED, the rate of CP in patients with acute pain was around 40%. Patients with CP come more frequently to ED than patients without CP. Their use of care structures, particularly ED, is all the more frequent that their disability is important. The satisfaction of these patients in ED is associated with age, nature of pain, wait duration, realisation of imaging, and administration of painkillers and relieving of pain. The reasons why these patients go to ED were pain exacerbation, inadequate strategy of coping, severity of disease and sometime despair associated with stress or anxiety. Currently the investigators do not know if these managements in ED are adequate or not. And finally the investigators do not know whether the satisfaction about their ED management is different from patients without CP. The investigators are going to collect data about all patients admitted in ED with the objective to compare the satisfaction between patients with CP and patients without CP. The follow up will be restricted to the area of ED. The last data will be collected just before the exit from ED.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more admitted in ED
* between 8 am and 5pm
* from Monday to Friday.

Exclusion Criteria:

* Patients admitted directly in emergency intensive care for vital distress defined by hemodynamic, respiratory, or neurological failure distress,
* multitrauma patients;
* patient without possibility to communicate because of neurologic disease or mental status disease;
* linguistic barrier.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study concerns emergency department population.
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-02-03 (Actual); Study Completion 2018-02-03 (Actual)

PRIMARY OUTCOMES:
Medical care modalities satisfaction | Day 1
  Proportion of patients satisfied or very satisfied with the management at the emergency department (ED)

SECONDARY OUTCOMES:
Rate of patients with chronic pain. | Day 1
  History of a chronic pain or daily pain since 3 months.
Duration of management between first medical contact and delivery from ED. | Day 1
  Time on arrival at the ED and time on discharge from ED.
Pain intensity | Day 1
  Measurement with numerical pain scale, from 0 (without pain) to 10 (the worst pain intensity imaginable).
Anxiety intensity | Day 1
  Measurement with numerical anxiety scale, from 0 (without anxiety) to 10 (the worst anxiety intensity imaginable).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pellegrin - Service des urgences adultes, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No